CLINICAL TRIAL: NCT06691646
Title: Effect of RECOGNeyes Training on Brain Networks
Brief Title: RECOGNeyes Gaze-Control Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Liddle, Associate Professor in Translational Mental Health, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CiC2017026
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Inattention; Cognitive Training; Cognitive Control; Oculomotor Dysfunction; Magnetoencephalography (MEG)
Keywords: gaze-control training; oculomotor control; attention deficit/hyperactivity disorder (ADHD); magnetoencephalography; dyslexia/reading disorder; resting state brain connectivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to undertake 2, 3 or 4 training sessions at home, per week, for 20 to 30 minutes per session over a period of two weeks. Total achieved training time is recorded and will be correlated with outcomes.
Who Masked: Outcomes Assessor
Masking Description: All researchers involved in data collection are masked until after data collection and preprocessing is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Two training sessions per week (Experimental): Train with RECOGNeyes gaze training game at home twice a week, for between 20 to 30 minutes per training session, for two weeks.
  Interventions: Behavioral: Gaze-control training game
- Three training sessions per week (Experimental): Train with RECOGNeyes gaze training game at home three times per week, for between 20 to 30 minutes per training session, for two weeks.
  Interventions: Behavioral: Gaze-control training game
- Four training sessions per week (Experimental): Train with RECOGNeyes gaze training game at home four times per week, for between 20 to 30 minutes per training session, for two weeks.
  Interventions: Behavioral: Gaze-control training game

INTERVENTIONS:
Behavioral: Gaze-control training game — An eyetracker-controlled computer game designed to improve attentional control by training inhibitory control over direction of gaze. It includes six mini-games, each designed to train different aspects of oculomotor control, including selective attention, motor inhibition, motor timing, and spatial working memory.
  Other Names: RECOGNeyes

SUMMARY:
RECOGNeyes is a computer game developed by members of the research team to improve attention in people who find it hard to "keep their eyes on the task". Players use a small eyetracker to control the game with their eyes, giving their gaze-control system (oculomotor control system) a thorough work-out.

This is a "confidence-in-concept" study to see whether RECOGNeyes holds promise as an approach to improving attentional control. It takes the form of a clinical trial, in which three groups of participants will undertake different amounts of RECOGNeyes training.

The goals of the study are to find out:

* Whether RECOGNeyes training changes patterns of brain activity during a challenging gaze-control task.
* What changes in brain activity participants show when their gaze control improves.

Before and after RECOGNeyes training, participants will have two kinds of brain scan:

1. Magnetoencephalography to measure their brain waves while they do a gaze-control task that involves shifting their gaze to look either towards, or away from, an object that suddenly appears on the left or right side of a screen. It takes extra control to look away from the object as they have to actively resist the strong impulse to look towards it.
2. Functional magnetic resonance imaging of the brain while the participants are at rest in the scanner, with their eyes open. This reveals the connection patterns between different parts of the brain when the participant is not doing anything in particular.

Participants will be healthy young adults, and recruitment will focus on young people who are receiving academic support for their studies, as they are more likely to have problems with "keeping their eyes on the task".

They will be given sealed written instructions to play RECOGNeyes at home two, three or four times per week for two weeks, playing for 20 to 30 minutes at a time. How many times per week they are to play will be decided by random draw.

From the scanning data, the researchers will:

* Measure changes in brain waves and brain connectivity before and after training.
* Measure improvements in the gaze-control task and how strongly the improvements relate to brain changes.
* See whether the brain changes relate to how long the participants spent training.

If participants who trained for longer show more improved gaze control, as well as greater brain changes, this will provide grounds for confidence in the RECOGNeyes approach to improving inattention.

DETAILED DESCRIPTION:
STUDY PURPOSE

RECOGNeyes is an eyetracker-controlled training game the researchers have developed in collaboration with young people with Attention Deficit/Hyperactivity Disorder (ADHD), their parents, and their teachers. It is designed to improve cognitive control in these conditions by training greater inhibitory top-down control over direction of gaze. The goal of this study is to establish whether there are grounds for confidence in the concept of gaze-control training as an approach to improving attentional control in conditions such as ADHD. The researchers will do this by investigating neural correlates of oculomotor control before and after RECOGNeyes gaze-control training, and evaluating the extent to which changes in these neural correlates themselves are associated with improved oculomotor control and with time spent training.

The researchers will use magnetoencephalography (MEG) recorded while participants undertake an antisaccade task, to evaluate electrophysiological correlates of oculomotor control. They will use resting state functional MRI to evaluate changes to functional connectivity between nodes of brain networks involved in visual attention and oculomotor control.

OBJECTIVES:

* To measure changes in electrophysiological event-related spectral perturbation (ERSPs) associated with topdown control of saccadic eye movements during an "antisaccade" task after participants have undertaken two weeks of RECOGNeyes training.
* To measure changes in resting state connectivity between brain regions involved in visual attention and oculomotor control.
* To correlate these neural changes with training gains (measured as improvements in antisaccade task performance) and with time spent training. Associations between neural changes and improved performance will indicate that improvements in oculomotor control are reflected in alterations to underlying neural function, while associations between time spent training, training gains, and neural changes will indicate that these changes are likely to reflect RECOGNeyes training effects.
* To explore the user experience of participating in the training and identify facilitators and barriers to using RECOGNeyes as a tool for gaze-control training.

PARTICIPANTS

The researchers plan to recruit at least 30 healthy volunteers from students accessing Academic Support Services at local further and higher education establishments in Nottingham. This strategy is designed to yield a sample of young adults that is enriched for inattentiveness. Posters and recruitment emails will be used to advertise the study. If the researchers are unable to recruit 30 volunteers from Academic Support Services, the researchers will also recruit from the general population by advertising more widely around the University of Nottingham.

The researchers will invite 8-12 of the participants to take part in qualitative interviews to explore their user experience with RECOGNeyes. Participants will be recruited for these interviews concurrently on completion of their follow-up scans, and recruitment for these interviews will cease upon data saturation.

STUDY DESIGN

Participants will attend the Sir Peter Mansfield Imaging Centre (SPMIC), University of Nottingham, on two occasions, before and after undertaking RECOGNeyes training at home over a period of two weeks. Over the training period, the researchers will provide the participants with a laptop computer on which the game is installed, together with a small USB eye-tracker that can be mounted under the laptop screen with a magnetic mount.

Each visit to SPMIC will include an MEG scan lasting approximately 40 minutes, during which they perform an antisaccade task; and a MRI scanning session that includes both an anatomical scan for co-registration with the MEG data to allow source localisation, and a short resting state functional scan (eyes open).

At the first visit only, after providing written consent to participate in the study, participants will complete the self-report Conners Adult ADHD Rating Scale (CAARS) (Conners et al. 1999). This will provide measures of the levels of inattention and hyperactivity/impulsivity in the participant sample. At both visits, participants will also complete two measures of reading efficiency: the TOWRE-2 standardised test of single word reading (Torgesen, 2011), which captures both word recognition efficiency using a list of real words, and phonetic decoding efficiency using a list of pseudo-words; and a custom task designed to measure eye-movement efficiency, in which they silently read three short passages of text while their eye movements are recorded. They will also, on both visits, complete the 12 item version of the General Health Questionnaire (GHQ12) (Goldberg & Williams, 1988), to assess their general mental health and to allow researchers to evaluate whether gaze-control training has had any impact on their mental wellbeing, whether positive or adverse.

The antisaccade task performed in the MEG scanner consists of 40 blocks of six trials. Twenty of these blocks are "prosaccade" blocks in which participants have to make a saccadic eye movement from a central fixation cross to a stimulus presented either to right or left of fixation. The other 20 blocks are "antisaccade" blocks, in which they have to make a counter-intuitive saccade in the opposite direction to the peripheral stimulus. Each stimulus is preceded by a warning cue 800ms earlier, to allow them to prepare to make their saccadic response. After their response is completed, they receive feedback as to whether their saccade was correct or incorrect, and whether it was made within the time limit. They are awarded a point for a timely saccade in the correct direction, and a point is deducted for an incorrect or late response. Block type order is randomised, and blocks are separated by rest periods.

For those recruited to participate in the qualitative interview, this takes place on a third visit to the University of Nottingham, and lasts approximately one hour.

RANDOMISATION AND BLINDING

Participants are randomly assigned to undertake two, three or four training sessions per week for two weeks (training sessions to last 20-30 minutes), at home. Randomisation will be stratified by age, gender and nature of academic difficulty (e.g. ADHD; dyslexia) on a rolling basis as volunteers are recruited. Training instructions will be given to volunteers in a sealed envelope, and investigators involved in pre- and post-intervention measurements will remain blind to training schedule allocation until after data have been processed (CAARS, reading, and GHQ12 measures scored; MEG, eye-tracker and fMRI data pre-processed).

This randomised scheduling protocol is designed to produce variability between participants in the amount of time spent training, so that changes in outcome measures before and after training can be correlated with actual time spent training, and thus provide the researchers with evidence as to whether training gains and/or neural changes observed after the two-week training period are attributable to RECOGNeyes training, rather than simply to greater familiarity with the outcome measure assessment procedures on the second visit.

The Chief Investigator (Dr. Elizabeth Liddle) will maintain a record of which volunteers have been allocated to which training schedule. Volunteers will be given her contact details so that if they experience any problem with their training or training schedule, they can to contact her directly for help.

TRAINING COMPLIANCE

The RECOGNeyes software installed on the laptops will log the time participants begin and end each training session, and will be used to quantify the actual training time achieved by each participant.

PARTICIPANT WITHDRAWAL

Participants may be withdrawn from the study either at their own request or at the discretion of the researchers. The participants will be made aware that this will not affect their future care. Participants who withdraw early in the study may be replaced.

DATA ANALYSIS PLAN

This study was designed, in accordance with the funding call (MRC Confidence in Concept), as an exploratory study to provide evidence that RECOGNeyes training can result in changes to brain networks involved in cognitive control. As an exploratory, proof-of-concept study, the study has not been powered to find effects of specified size. Instead, the researchers will look at a range of possible indicators of the impact of RECOGNeyes training on cognitive control capacity, with a hierarchy of hypothesised effects to test for. Using MEG, Hwang et al.(2014) have shown that when participants prepare to make an antisaccade, oscillatory activity associated with functional inhibition increases in a brain region associated with top-down control (right dorsolateral prefrontal cortex), and is causally coupled with oscillatory activity in the frontal eye-fields, brain regions implicated in saccade generation. In a later study, Hwang et al. (2016) also demonstrated that these oscillatory correlates of top-down saccadic control develop over adolescence, suggesting that they may index cognitive control capacity, and, specifically, capacity to control direction of gaze. If RECOGNeyes training is successful in modulating this capacity, training gains should be correlated with changes in these correlates of top-down saccadic control. Therefore, the researchers plan to test for linear correlations between both training gains, as measured by antisaccade task performance, and/or training exposure (time actually spent training, calculated from game logs), and changes on our outcome measures.

The qualitative data gained from Day 3 will be analysed using thematic analysis (Braun & Clarke, 2006). This is a flexible approach that allows for the integration of both a deductive and inductive lens upon the data, enabling a combination of both theoretical views already known to the researchers, and the emergence of new themes introduced by the participants. Data will be managed using a framework approach, allowing for comparisons and contrasts to be drawn between and across cases in the data set.

ADVERSE EVENTS

Adverse events as a result of RECOGNeyes training are not expected. The research MRI scan is not the same as a routine clinical scan and therefore cannot be used to make a clinical diagnosis. However, there is a small chance of an incidental finding of potential clinical significance. This chance will be made known to participants as part of the consent process. The SPMIC has a standard operating procedure for such occurrences. If any scans reveal anything that suggests a possible clinical abnormality, the researchers will notify the participant's GP so that he or she can arrange any further investigations that might be indicated.

PUBLICATION AND DISSEMINATION

Results from this study will be published in academic journals. Participants will be informed that they may request copies of any published articles related to this study and that they will not be identified in any report or publication.

USER AND PUBLIC INVOLVEMENT

The RECOGNeyes gaze-control training programme and study design were developed in close collaboration with Patient and Public Involvement (PPI) groups.

FUNDING

This study is funded by the University of Nottingham via the Medical Research Council (MRC) Confidence-in-Concept (CiC) awards.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-30 years
2. Ability to give informed consent
3. We will prioritise recruiting volunteers who have ADHD, dyslexia, dyspraxia or dyscalculia
4. Normal or corrected-to-normal vision

Exclusion Criteria:

1. Magnetic Resonance Imaging safety exclusions
2. Partial sight or visual field deficit

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change in strength of alpha-beta oscillatory coupling | From enrolment day visit to second visit following two weeks gaze-control training.
  Change in strength of coupling between beta amplitude in right dorsolateral prefrontal cortex and high alpha amplitude in frontal eyefields during the cue-target period on anti-saccade trials, relative to prosaccade trials.
Change in beta-band oscillatory amplitude in dorsolateral pre-frontal cortex | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in beta-band (13-30 Hz) ERSP during the cue-target period of anti-saccade trials, relative to prosaccade trials.
Changes in alpha-band oscillatory amplitude in frontal eyefields | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in alpha-band (8-12 hz) ERSP during the cue-target period on anti-saccade trials, relative to prosaccade trials.

SECONDARY OUTCOMES:
Changes in degree of post-stimulus beta desynchronisation and synchronisation | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in post-stimulus beta desynchronization and synchronisation in attentional network nodes (frontal eyefields, dorsolateral prefrontal cortex, anterior insula, parietal eyefields; primary visual cortex) on antisaccade relative to prosaccade trials.
Changes in antisaccade task performance | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in performance on the anti-saccade task, as measured by saccade latencies and directional accuracy on antisaccade relative to prosaccade trials.
Changes in event-related pupil dilation and vergence rates | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in pupil dilation rate and convergence rate (rate of decrease in the angle between the direction of gaze of each eye) between cue onset and saccadic response for anti-saccade trials, relative to prosaccade trials.
Changes in tonic pupil diameter and vergence | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in mean baseline (prior to cue onset) measures of pupil diameter and vergence angle for antisaccade vs prosaccade trial blocks.
Changes in single word reading efficiency | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in standardised scores of real-word reading and pseudo-word reading on the TOWRE-2 reading efficiency test.

OTHER OUTCOMES:
Changes in eye-movment patterns during reading | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in eye-movement patterns recorded during silent reading of passages of text. Standard eyemovement reading metrics will be used, including fixation duration, proportion of regressive saccades, preferred landing position and length of skipped words.
Changes in resting state brain connectivity | From enrolment day visit to second visit following two weeks gaze-control training.
  Changes in resting state brain connectivity as measured by correlations between Blood Oxygen Level Dependency (BOLD) signal timecourses recorded using fMRI from nodes of visual attention/oculomotor networks.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Liddle, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Faculty of Medicine and Health Sciences, University of Nottingham, Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At the time of the study start, the implications of new data protection legislation was unclear, and protocols for IDP anonymisation were still being developed.

REFERENCES:
- [Background] Braun V, Clarke, V:Using thematic analysis in psychology. Qualitative Research in Psychology. 2006 3:2, 77-101.
- [Background] Hwang K, Ghuman AS, Manoach DS, Jones SR, Luna B. Frontal preparatory neural oscillations associated with cognitive control: A developmental study comparing young adults and adolescents. Neuroimage. 2016 Aug 1;136:139-48. doi: 10.1016/j.neuroimage.2016.05.017. Epub 2016 May 10. PMID 27173759
- [Background] Hwang K, Ghuman AS, Manoach DS, Jones SR, Luna B. Cortical neurodynamics of inhibitory control. J Neurosci. 2014 Jul 16;34(29):9551-61. doi: 10.1523/JNEUROSCI.4889-13.2014. PMID 25031398
- [Background] Goldberg DP, Williams P: A user's guide to the General Health Questionnaire. 1988, Basingstoke NFER-Nelson
- [Background] Conners CK, Ehrhard D, Sparrow D. CAARS Adult ADHD Rating Scales. New York: Multi-Health Systems; 1999.